CLINICAL TRIAL: NCT02818205
Title: Electrodermal Patterns of Arousal in Children With Autism Spectrum Disorder
Brief Title: Electrodermal Patterns of Arousal in Children
Status: Completed | Type: Observational
Sponsor: Barpak Geriatric Health Services, Inc. d/b/a Barpak Occupational Therapy (Other)
Responsible Party: Sponsor
Other Study IDs: Barpak-02-EDA
Record Dates: First submitted 2016-06-20; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children with Autism Spectrum Disorder: Boys between the age of 4 to 11 years old with Autism Spectrum disorder will participate in the Sensory Challenge Protocol which will measure electrodermal activity in response to sensation
  Interventions: Other: Sensory Challenge Protocol
- Typically Developing Children: Typically developing boys between the age of 4 to 11 years will participate in the Sensory Challenge Protocol which will measure electrodermal activity in response to sensation.
  Interventions: Other: Sensory Challenge Protocol

INTERVENTIONS:
Other: Sensory Challenge Protocol — Measurement of electrodermal activity in response to sensation

SUMMARY:
The purpose of this study was to explore the feasibility of detecting physiological patterns of arousal to sensory inputs in children with and without Autism Spectrum Disorder (ASD). Accordingly, two questions directed this methodological research investigation: (1) Is there a relationship between rest (tonic) and response (phasic) patterns of arousal among typically developing children and children with ASD?, and (2) Is there a difference in EDA response to sensation between typically developing children and children with ASD?

DETAILED DESCRIPTION:
This methodological research design is a prospective exploratory test-retest design assessing the relationship between tonic and phasic Electrodermal Activity (EDA) variables. EDA during rest and in response to a variety of sensations was measured using skin conductance. Descriptive statistics summarized EDA dependent variable data using skin conductance response (SCR) magnitude, SCR amplitude, skin conductance level (SCL), non-specific response (NSR) and habituation (HAB). The data was used to assess the relationship between tonic and phasic patterns of arousal and compare response patterns between groups using the Sensory Challenge Protocol (SCP) in children with ASD and typically developing children (TD).

ELIGIBILITY:
Inclusion Criteria: Boys ages 4 - 11 years old.

* Able to sit for 30 minutes and follow simple directions.
* Children with confirmed Autism Spectrum Disorder via School records or parent report.
* Typically developing children free of medical or neurological conditions.

Exclusion Criteria:

* Medical or neurological conditions other than Autism.
* Hearing loss or visual impairments.
* Children taking medications known to affect arousal.
* Children who are not able to follow simple commands.

Ages: 4 Years to 11 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A convenience sample of boys between the ages of 4 - 11 years with and without a diagnosis of Autism Spectrum Disorder were recruited from private and public New Jersey Schools, Barpak Occupational Therapy clinic, Bergenfield, New Jersey and Seton Hall University campus.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Electrodermal Activity in response to sensation: tonic and phasic skin conductance in MicroSiemens | Within six weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LACEY JI, LACEY BC. The relationship of resting autonomic activity to motor impulsivity. Res Publ Assoc Res Nerv Ment Dis. 1958;36:144-209. No abstract available. PMID 13527784
- [Background] MUNDY-CASTLE AC, MCKIEVER BL. The psychophysiological significance of the galvanic skin response. J Exp Psychol. 1953 Jul;46(1):15-24. doi: 10.1037/h0060100. No abstract available. PMID 13069662
- [Background] Schell AM, Dawson ME, Filion DL. Psychophysiological correlates of electrodermal lability. Psychophysiology. 1988 Nov;25(6):619-32. doi: 10.1111/j.1469-8986.1988.tb01899.x. No abstract available. PMID 3241850
- [Background] Schoen SA, Miller LJ, Brett-Green BA, Nielsen DM. Physiological and behavioral differences in sensory processing: a comparison of children with autism spectrum disorder and sensory modulation disorder. Front Integr Neurosci. 2009 Nov 3;3:29. doi: 10.3389/neuro.07.029.2009. eCollection 2009. PMID 19915733
- [Background] Vetrugno R, Liguori R, Cortelli P, Montagna P. Sympathetic skin response: basic mechanisms and clinical applications. Clin Auton Res. 2003 Aug;13(4):256-70. doi: 10.1007/s10286-003-0107-5. PMID 12955550